CLINICAL TRIAL: NCT03535909
Title: Hemodynamic Assessment Throughout Diuretic Treatment in Acute Decompensated Heart Failure
Brief Title: Hemodynamic Assessment in Acute Decompensated Heart Failure
Status: Completed | Type: Observational
Sponsor: Rodin Scientific LLC (Industry)
Collaborators: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RS-2018-S01
Record Dates: First submitted 2018-04-16; First posted 2018-05-24 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Congestive Heart Failure
Keywords: CHF; central venous pressure; noninvasive; ADHF; stroke volume
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Noninvasive Hemodynamic Measurement System — Ability of the noninvasive hemodynamic measurement system to determine changes in the hemodynamic status of heart failure patients admitted to the hospital with a primary diagnosis of acute decompensated heart failure.

SUMMARY:
This study will assess the ability of a novel optical measurement system to determine changes in the hemodynamic status of heart failure patients admitted to the hospital with a primary diagnosis of acute decompensated heart failure. Patients will be measured with both the novel measurement system and reference devices that are FDA-cleared for hemodynamic measurements. The measurements from the novel system will be compared to reference variables describing hemodynamic and congestive status, including stroke volume, central venous pressure, and serum levels of NT-proBNP.

DETAILED DESCRIPTION:
This study will assess the ability of a novel optical measurement system to determine changes in the hemodynamic status of heart failure patients admitted to the hospital with a primary diagnosis of acute decompensated heart failure. Patients will be measured with both the novel measurement system and reference devices that are FDA-cleared for hemodynamic measurements. The measurements from the novel system will be compared to reference variables describing hemodynamic and congestive status, including stroke volume, central venous pressure, and serum levels of NT-proBNP.

All patients enrolled in the study will first provide written informed consent to participate and then the research coordinator will check that the subject meets all study inclusion criteria and does not meet any of the study exclusion criteria. Enrolled subjects will undergo up to six (6) hemodynamic assessment sessions lasting less than 90 minutes each over the course of their hospitalization. There will be at least eight (8) hours between assessment sessions.

Each assessment session includes recording of the subject's weight, measurements with the reference devices, and measurements with the novel optical system. During the session, the subject will be assessed in the supine, sitting, and standing positions. NT-proBNP measurements will be done at the start of study participation and the end. A market research questionnaire will be administered to the subject following the first measurement session.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to the hospital with a primary diagnosis of acute decompensated heart failure
* Treated with or planned treatment with intravenous diuretics
* Volume overload, as indicated by at least one of the following clinical signs:

  * Peripheral edema
  * Pulmonary edema on physical examination
  * Pleural effusions on chest x-ray
  * Jugular venous distension on physical examination
  * CVP > 10 cmH2O
  * Presence of third heart sound
* Able to understand study procedures, agree to participate in the study program and voluntarily provide written informed consent

Exclusion Criteria:

* Inability or refusal to sign the Subject Informed Consent
* Age > 80 years
* Body mass index (BMI) > 40
* Planned mechanical ventilation during hospitalization
* Presence of left ventricular assist device (LVAD)
* Dialysis
* Pregnancy. All women of childbearing potential must have a negative pregnancy test before enrollment.
* Parenteral diuretic or other medical treatment for ADHF already administered for more than 12 hours prior to enrollment
* Skin damage to the optical sampling sites (fingers and dorsal hand), to include tattoos, scars, cuts, or burns extending over more than 30% of the visible tissue
* Compromised superficial hand veins or proximal venous stenosis
* Intravenous lines connected to both arms
* Inability to stand with support, if needed, for 4 minutes
* Inability to place hand in the venous imaging enclosure due to forearm, elbow, or shoulder injuries, or other physical constraints
* Inability to wear fingertip or ring sensors on three fingers (of either hand) due to missing fingers, injured fingers, or other physical constraints
* Persons in police custody or prisoners
* Major medical or psychiatric condition that would interfere with the ability to complete the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with congestive heart failure and admitted to the hospital with a diagnosis of acute decompensated heart failure (ADHF).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-06-09 (Actual); Primary Completion 2018-06-24 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of Estimated Changes in Stroke Volume | Retrospective up to 6 months after study completion
  Comparison of Stroke Volume Measurement (units of ml) from the optical measurement system with paired Stroke Volume Measurement (ml) from the reference device. Accuracy will be measured in percentage error and Bland-Altman limits of agreement.

SECONDARY OUTCOMES:
Accuracy of Central Venous Pressure Measurement | Retrospective up to 6 months after study completion
  Comparison of Central Venous Pressure Measurement (units of cmH2O) from the optical measurement system with paired Central Venous Pressure Measurement (cmH2O) from the reference device. Accuracy will be measured in percentage error and Bland-Altman limits of agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Allen, PhD, Principal Investigator — Rodin Scientific
Locations (2):
- New Mexico Heart Institute, Albuquerque, New Mexico, United States
- University Hospital of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No